CLINICAL TRIAL: NCT01799525
Title: Therapeutical Hypercapnia to Prevent Secondary Ischemic Events in Aneurysmal Subarachnoid Hemorrhage (aSAH)
Brief Title: Hypercapnia to Prevent Secondary Ischemia in SAH
Acronym: SAHCO2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Principal Investigator, Dr. Thomas Westermaier, MD, Wuerzburg University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: WUE102/12
Record Dates: First submitted 2013-02-20; First posted 2013-02-26 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage
Keywords: Aneurysm; subarachnoid hemorrhage; vasospasm; cerebral ischemia; stroke
MeSH Terms: conditions — Subarachnoid Hemorrhage; Aneurysm; Brain Ischemia; Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hypercapnia (Experimental): Intervention: SAH patients are subjected to gradual hypercapnia by reduction of respiratory volume in one trial session every day. PaCO2 is raised from normocapnia to 50 mmHg for 10 - 15 minutes and 60 mmHg for 10 - 15 minutes.
  Interventions: Procedure: Hypercapnia by reduction of respiratory volume

INTERVENTIONS:
Procedure: Hypercapnia by reduction of respiratory volume — By reduction of the respiratory volume, PaCO2 is raised while paO2 is kept constant by modulation of the oxygen supply through the respirator,

SUMMARY:
Delayed cerebral vasospasm and secondary ischemic infarction are feared complications after aneurysmal subarachnoid hemorrhage (aSAH). To date, there is no effective therapy to prevent these ischemic complications. The arterial partial pressure of carbon dioxide (PaCO2) is one of the main determinants of cerebral blood flow (CBF) in healthy subjects. It is yet largely unknown, if and to what extent modulations of PaCO2 can influence CBF in patients after aSAH. The trial is a phase 1 study in which the feasibility of hypercapnia in SAH patients is tested. PaCO2 is gradually raised to 60 mmHg in 10 mechanically ventilated aSAH patients. Cerebral oxygen saturation measured by NIRS and CBF determined by an intracerebral thermodilution probe are the primary end points. If the feasibility is confirmed, this trial will be followed by a phase 2 dose finding study.

DETAILED DESCRIPTION:
The course of aneurysmal subarachnoid hemorrhage (aSAH) is determined by the sequence of several ischemic episodes. Immediately after aSAH, an increase of ICP causes an increase of CBF. It is followed by an acute vasoconstriction over the next hours and days. Typically between day 4 and 10 after aSAH, delayed arterial narrowing and a decrease of CBF occurs in approximately 50 % of aSAH patients and may result in cerebral ischemia and infarction. After the failure of the CONSCIOUS-trial to improve outcome after aSAH, there is no specific treatment in sight to effectively prevent cerebral ischemic events after aSAH. Under physiological conditions, the arterial partial pressure of carbon dioxide (PaCO2) is one of the main determinants of cerebral blood flow (CBF). An elevation of PaCO2 may also be a useful treatment on aSAH patients. This trial is designed as a phase 1 study to test the feasibility of controlled hypercapnia in mechanically ventilated aSAH patients with poor-grade SAH. Monitoring is performed by an external ventricular drainage (ICP), near infrared spectroscopy (tissue oxygenation) and a thermodilution probe (CBF). The latter monitoring tools represent the primary end points of this study. In case of affirmed feasibility, a dose finding study will be launched as a next step.

ELIGIBILITY:
Inclusion Criteria:

* aneurysmal SAH
* SAH Hunt/Hess Grade 3-5
* SAH Fisher Grade 2-4
* Mechanically ventilated
* external ventricular drainage/ICP measurement

Exclusion Criteria:

* Age under 18
* ICP > 25 mmHg for > 2 minutes
* pH < 7.250

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-01; Primary Completion 2014-02 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Cerebral Blood Flow | For an average of two weeks after aSAH
  Between day 4 and 14, PaCO2 is gradually raised from normocapnic values (40 mmHg) to hypercapnic values (50 and 60 mmHg). CBF is continuously measured during this intervention. Patients are clinically and radiologically followed for 6 months.

SECONDARY OUTCOMES:
Cerebral oxygen saturation | For an average of two weeks after aSAH
  Oxygen saturation by NIRS is measured continuously for 2 weeks after aSAH.
intracranial pressure (ICP) | For an average of two weeks
  ICP is continuously measured by an external ventricular drainage throughout the intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Westermaier, MD, Principal Investigator — Department of Neurosurgery, University of Wuerzburg, Germany; Ekkehard Kunze, MD, Study Director — Department of Neurosurgery, University of Wuerzburg
Locations (1):
- Department of Neurosurgery, University of Wuerzburg, Würzburg, Bavaria, Germany

REFERENCES:
- [Derived] Stetter C, Weidner F, Lilla N, Weiland J, Kunze E, Ernestus RI, Muellenbach RM, Westermaier T. Therapeutic hypercapnia for prevention of secondary ischemia after severe subarachnoid hemorrhage: physiological responses to continuous hypercapnia. Sci Rep. 2021 Jun 3;11(1):11715. doi: 10.1038/s41598-021-91007-7. PMID 34083595
- [Derived] Westermaier T, Stetter C, Kunze E, Willner N, Holzmeier J, Kilgenstein C, Lee JY, Ernestus RI, Roewer N, Muellenbach RM. Controlled transient hypercapnia: a novel approach for the treatment of delayed cerebral ischemia after subarachnoid hemorrhage? J Neurosurg. 2014 Nov;121(5):1056-62. doi: 10.3171/2014.7.JNS132611. Epub 2014 Aug 22. PMID 25148012